CLINICAL TRIAL: NCT03657186
Title: Double-blind, Randomised, Placebo-controlled Study to Evaluate Benefit of ProbioSatys™ on Weight Reduction in Overweight Subjects
Brief Title: Study to Evaluate Benefit of ProbioSatys™ on Weight Reduction in Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TargEDys (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAR/006118
Record Dates: First submitted 2018-08-02; First posted 2018-09-04 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Overweight; Weight Loss
Keywords: Probiotics; Microbiome; Microbiota; Hafnia alvei; Overweight; Food intake; Appetite regulation; Satiety; Weight loss; Glucose Metabolism; Glycemia; Enterobacteriaceae; Gut-brain axis; Molecular mimicry
MeSH Terms: conditions — Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProbioSatys™ (Experimental)
  Interventions: Dietary Supplement: ProbioSatys™
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: ProbioSatys™ — One capsule, twice a day, is to be orally taken with 100 mL of water during each breakfast and lunch (approx. 5 minutes after starting eating), total 2 capsules per day.
  Arms: ProbioSatys™
Other: Placebo — One capsule, twice a day, is to be orally taken with 100 mL of water during each breakfast and lunch (approx. 5 minutes after starting eating), total 2 capsules per day.
  Arms: Placebo

SUMMARY:
The study aims to evaluate the effects of ProbioSatys™ on body weight and related parameters in overweight subjects during a 12-week consumption period. In addition, tolerability and safety of ProbioSatys™ will be assessed.

DETAILED DESCRIPTION:
ProbioSatys™ is a probiotic nutritional solution containing a commensal Enterobacteriaceae food grade strain, Hafnia alvei 4597. The microbiome is known to play a crucial role in body weight management and metabolic disease. ProbioSatys™ mechanism of action relies on bacterial metabolites that send local and central signals via the gut-brain axis by molecularly mimicking satiety hormones involved in appetite regulation.

Numerous ProbioSatys™pre-clinical studies indicate that consumption of the strain leads to body weight loss based on food intake reduction, but also improvement of body composition (increase of lean mass/fat mass ratio), and improvement of glucose metabolism (oral glucose tolerance test, and fasted glycemia).

The present study aims to evaluate the effects of ProbioSatys™ on body weight and related parameters in overweight subjects during a 12-week consumption period. In addition, tolerability and safety of ProbioSatys™ will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old males and females
2. Overweight (Body Mass Index, BMI: 25 kg/m2 - 29.9 kg/m2)
3. Generally in good health
4. Desire to lose weight
5. Regularly consuming 3 main meals/day (breakfast, lunch, dinner)
6. Readiness to comply with study procedures, in particular:

   * Follow diet recommendation
   * Maintain the habitual level of physical activity during the study
   * Fill out the questionnaires and subject diary
   * Take the IP as instructed
7. Stable body weight in the last 3 months prior to V1 (≤5% self-reported change)
8. Stable concomitant medications (if any) for at least last 3 months prior to V1
9. Women of childbearing potential:

   * Negative pregnancy testing (beta HCG-test in urine) at V1
   * Women of childbearing potential: commitment to use contraception methods (with the exception of starting new contraception medication)

Participation is based upon written informed consent form by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Randomisation criteria (to be checked after run-in at V2):

1. No change in body weight or reduction up to 3 kg (compared to V1)
2. Adequately completed subject diary
3. Readiness and ability to comply with study requirements
4. Relevant inclusion and exclusion criteria met

Exclusion Criteria:

1. Known allergy/sensitivity to any components of the investigational product
2. Pathological electrocardiogram (ECG) at V1
3. History and/or presence of clinically significant self-reported disorder as per investigator's judgement:

   * Untreated or non-stabilised thyroid gland disorder
   * Untreated or non-stabilised hypertension (regular systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg)
   * Digestion/absorption disorders of the gastrointestinal tract (e.g. inflammatory bowel disease, coeliac disease, pancreatitis etc.) and/ or gastrointestinal surgery
   * Diabetes mellitus type 1 or untreated/non-stabilised type 2
   * Acute or chronic psychotic disorder
   * Immunodeficiency
   * Any other organ or systemic diseases that could influence the conduct and/or outcome of the study and/or could affect the tolerability of the subject
4. History and/or presence of eating disorders like bulimia, anorexia nervosa, binge-eating as per investigator's judgement
5. Any electronic medical implant
6. Deviation of safety laboratory parameter(s) at V1 that is:

   * Clinically significant or
   * >2x upper limit of normal, unless the deviation is justified by a previously known not clinically relevant condition (e.g. Gilbert's syndrome)
7. Use of medication/supplementation in the last month prior to V1 and during the study, as per investigator's judgement:

   * That could influence gastrointestinal functions (such as antibiotics, probiotics, laxatives, opioids, anticholinergics, anti-diarrheals etc.)
   * For weight management (e.g. fat binder/burner, satiety products etc.)
   * That could influence body weight (e.g. antidepressants, systemic corticoids etc.)
   * That could otherwise interfere with study conduct / evaluation
8. Diet/weight loss programs within the last 3 months prior to V1 and during the study
9. Smoking cessation/modification of smoking level (if any) within 6 months prior to V1 and/or during the study (regular smoking during the study at the same level as prior to the study is allowed)
10. Vegetarian, vegan or other restrictive diet
11. Pregnancy or nursing
12. History of or current abuse of drugs, alcohol or medication
13. Inability to comply with study procedures
14. Participation in another study during the last 30 days prior to V1
15. Any other reason deemed suitable for exclusion, per investigator's judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who lost at least 3% of baseline body weight (="3% responders") | 12 weeks

SECONDARY OUTCOMES:
Body weight change (in kg), compared to baseline (V2) | 4, 8 and 12 weeks
Body weight change (%), compared to baseline (V2) | 4, 8 and 12 weeks
Body weight (in kg ) | 4, 8 and 12 weeks
Proportion of subjects who lost at least 3% of baseline body weight (="3% responders") | 4 and 8 weeks
Proportion of subjects who lost at least 5% of baseline body weight (="5% responders") | 4, 8 and 12 weeks
Body fat mass assessed per bioelectrical impedance analysis (BIA), compared to baseline | 4, 8 and 12 weeks
Body fat free mass assessed per bioelectrical impedance analysis (BIA), compared to baseline | 4, 8 and 12 weeks
Waist circumference, compared to baseline | 4, 8 and 12 weeks
Hip circumference, compared to baseline | 4, 8 and 12 weeks
Lipid metabolism parameters (total cholesterol), compared to screening values (V1) | 14 weeks
Lipid metabolism parameters (high density lipid cholesterol), compared to screening values (V1) | 14 weeks
Lipid metabolism parameters (low density lipid cholesterol), compared to screening values (V1) | 14 weeks
Fasting glucose, compared to screening values (V1) | 14 weeks
Glycated haemoglobin (HbA1c), compared to screening values (V1) | 14 weeks
Evaluation of the overall feeling of satiety compared to baseline by using visual analogue scales (VAS) | 4, 8 and 12 weeks
  continuous line between two endpoints: not saturated at all & fully saturated
Evaluation of the overall feeling of fullness compared to baseline by using visual analogue scales (VAS) | 4, 8 and 12 weeks
  continuous line between two endpoints: not full at all & extremely full
Evaluation of the overall feeling of craving compared to baseline by using a 5 point Likert scale | 4, 8 and 12 weeks
  0= "no", 1= "slightly", 2= "moderate", 3= "strong" and 4= "very strong"
General well-being parameters (Impact of Weight on Quality of Life-Lite, IWQOL-LITE), compared to baseline | 4, 8 and 12 weeks
Global evaluation of benefit at V5 by subject and the investigator | 12 weeks
  "very good", "good", "moderate" and "poor"

OTHER OUTCOMES:
Assessment of adverse events throughout the study | 14 weeks
Blood pressure, compared to baseline | 4, 8 and 12 weeks
Pulse rate, compared to baseline | 4, 8 and 12 weeks
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  analysis of full blood count parameters (haemoglobin)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  analysis of full blood count parameters (haematocrit)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  analysis of full blood count parameters (thrombocytes)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  analysis of full blood count parameters (leucocytes)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  liver and renal function parameters (alanine transaminase)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  liver and renal function parameters (aspartate aminotransferase)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  liver and renal function parameters (gamma-glutamyltransferase)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  liver and renal function parameters (alkaline phosphatase)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  liver and renal function parameters (bilirubin)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  liver and renal function parameters (creatinine)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  liver and renal function parameters (urea)
Safety laboratory parameters, compared to screening values (V1) | 14 weeks
  liver and renal function parameters (uric acid)
Global evaluation of tolerability at V5 by subject and the investigator | 12 weeks
  "very good", "good", "moderate" and "poor"
Gastrointestinal tolerability parameters (Gastrointestinal Symptom Rating Scale questionnaire, GSRS), compared to baseline | 4, 8 and 12 weeks
Stool frequency in the week before each visit post- baseline, each compared to the week before baseline (V2) | 4, 8 and 12 weeks
Physical activity parameters (Global Physical Activity Questionnaire, GPAQ), compared to baseline | 4, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Analyze & Realize, Berlin
  - Barbara Grube, Berlin
  - Jörg Förstermann, Berlin

IPD SHARING:
Plan to Share IPD: No